CLINICAL TRIAL: NCT04497441
Title: Perceptions of Netizens Regarding COVID-19 Information & Information Sources: A Cross Sectional Study
Brief Title: Netizens' Perception of COVID-19 Information & Information Sources.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Dr Shiva Shankar Bugude, Assistant Professor, Qassim University
Other Study IDs: QassimU3
Record Dates: First submitted 2020-08-01; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Covid19; Information Seeking Behavior; Social Media; Perception, Self
Keywords: COVID-19; Information; Information sources; Netizens; Perception; Social media
MeSH Terms: conditions — COVID-19; Information Seeking Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Netizens: Internet users in Al Qassim province region are the target study population for this study. This Cross sectional study utilizes an electronic google form to get responses from netizens of Al Qassim province of Saudi Arabia regarding the perception of COVID-19 information and information sources. All the questions in the survey are compulsory answerable questions. The settings in the google form are set so that a single respondent can limit the survey response to single time. The Google form link is shared to the netizens of Al Qassim province across relevant Social media platforms.
  Interventions: Other: Electronic Survey questionnaire

INTERVENTIONS:
Other: Electronic Survey questionnaire — This Cross sectional study utilizes an electronic google form to get responses from netizens of Al Qassim province of Saudi Arabia regarding the perception of COVID-19 information and information sources. All the questions in the survey are compulsory answerable questions. The settings in the google form are set so that a single respondent can limit the survey response to single time. The Survey Questionnaire contained following sections:
  Section I: Minimum required personal details Section II: 10 Questions regarding the source of COVID-19 information Section III: 6 Questions regarding perception of the COVID-19 information
  The very first part of the Questionnaires seeks responders' consent for giving responses to the survey questions. participation Section II & III contained all closed ended questions. The Google form link is shared to the netizens of Al Qassim province across relevant Social media platforms.

SUMMARY:
COVID-19 Infection was characterized as a Pandemic by WHO on the 11th of March 2020.1 After this there were all possible worldwide efforts to increase awareness in the general population about the COVID-19 Infection signs, symptoms, mode of transmission and prevention. The information was spread across all possible mass media communication channels. There were constant updates regarding the data of newly infected cases, deaths, and recoveries. This cross sectional study is conducted with the following objectives:

1. To understand the netizens perception regarding the sources of information available on COVID-19.
2. To understand the netizens populations perception regarding the available information on COVID-19.

DETAILED DESCRIPTION:
Mass media plays a significant role in public outreach and create awareness. Various mass media has their individual reach to the general public. In the current world of information technology availability of information is not an issue. There is in fact excessive availability of information. What makes a big difference is that RIGHT information delivery on RIGHT time and within RIGHT time. After WHO characterized COVID-19 infection as pandemic, mass media played a significant role in creating awareness regarding COVID-19 infection signs, symptoms, mode of transmission and its prevention. There were constant updates in various mass media regarding the data of newly infected cases, deaths, and recoveries. COVID-19 Pandemic has created fears, anxiety, and worries among the general population. There was information given to general public regarding treatment drugs and possibility of vaccine for COVID-19 infection. This created a ray of hope in many. So information in various mass media sources had different types of impact on general population thoughts.

This cross sectional study is conducted with the following objectives:

1. To understand the general populations perception regarding the sources of information available on COVID-19.
2. To understand the general populations perception regarding the available information on COVID-19.

This Cross sectional study utilizes an electronic google form to get responses from netizens of Al Qassim province of Saudi Arabia regarding the perception of COVID-19 information and information sources. All the questions in the survey are compulsory answerable questions. The settings in the google form are set so that a single respondent can limit the survey response to single time. The Survey Questionnaire contained following sections:

Section I: Minimum required personal details Section II: 10 Questions regarding the source of COVID-19 information Section III: 6 Questions regarding perception of the COVID-19 information

The questionnaire also carried the following disclaimer:

"This Survey will not Collect your Name, Email, Location, and Phone number. We pledge that the data obtained by this survey is for Educational purpose & scientific knowledge enhancement only. The data will not be transferred or shared with any other third party for commercial interest."

The very first part of the Questionnaires seeks responders' consent for giving responses to the survey questions. participation Section II & III contained all closed ended questions. The Google form link is shared to the netizens of Al Qassim province across relevant Social media platforms.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female Human volunteer internet users who belong &/or reside in Al Qassim province region of Saudi Arabia.
* Volunteers should be major by age (18 years and above).

Exclusion Criteria:

* Minor age group (<18 years) subjects are excluded from the study.
* Internet users who have preexisting phobia and/or anxiety mental conditions are excluded from the study.
* Internet users who are currently under treatment for their preexisting phobia and/or anxiety mental conditions are excluded from the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This online Observational Cross-sectional survey study is conducted to get responses from the Al Qassim province region Internet users. They are the target study population for this study. The Google form questionnaire survey link will be shared with the Dentists in internet via Social Media &/Or email to seek responses. The link will be available for single response for a single respondent.
Sampling Method: Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-08-10 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Netizens' perception of the Sources of COVID-19 information | 11th of August 2020
  Assessing the perception regarding the Sources of COVID-19 information among netizens in Al Qassim province using a 10 open ended Questionnaire. Descriptive statistics will be used to present the data.
Netizens' perception on COVID-19 information | 11th of August 2020
  Assessing the perception regarding COVID-19 information among netizens in Al Qassim province using a 6 open ended Questionnaire. Descriptive statistics will be used to present the data.

SECONDARY OUTCOMES:
Correlation of Age and the Frequency of checking COVID-19 information updates | 11th of August 2020
  The survey data will be statistically analyzed to check for the Correlation of Age and the Frequency of checking COVID-19 information updates. The data obtained from the survey will be subjected to appropriate analytical statistical tests to understand the correlation. A p-value of <0.05 is considered statistically significant correlation of the variables analysed.
Correlation of Gender and the Frequency of checking COVID-19 information updates | 11th of August 2020
  The survey data will be statistically analyzed to check for the Correlation of Gender and the Frequency of checking COVID-19 information updates. The data obtained from the survey will be subjected to appropriate analytical statistical tests to understand the correlation. A p-value of <0.05 is considered statistically significant correlation of the variables analysed.
Correlation of Age and the perception of newly infected COVID-19 cases information update | 11th of August 2020
  The survey data will be statistically analyzed to check for the Correlation of Age and the perception of newly infected COVID-19 cases information update. The data obtained from the survey will be subjected to appropriate analytical statistical tests to understand the correlation. A p-value of <0.05 is considered statistically significant correlation of the variables analysed.
Correlation of Age and the perception of COVID-19 deaths information update | 11th of August 2020
  The survey data will be statistically analyzed to check for the Correlation of Age and the perception of COVID-19 deaths information update. The data obtained from the survey will be subjected to appropriate analytical statistical tests to understand the correlation. A p-value of <0.05 is considered statistically significant correlation of the variables analysed.
Correlation of Age and the perception of COVID-19 Vaccine information update | 11th of August 2020
  The survey data will be statistically analyzed to check for the Correlation of Age and the perception of COVID-19 Vaccine information update. The data obtained from the survey will be subjected to appropriate analytical statistical tests to understand the correlation. A p-value of <0.05 is considered statistically significant correlation of the variables analysed.
Correlation of Age and the perception of COVID-19 treatment medicines/drugs information update | 11th of August 2020
  The survey data will be statistically analyzed to check for the Correlation of Age and the perception of COVID-19 treatment medicines/drugs information update. The data obtained from the survey will be subjected to appropriate analytical statistical tests to understand the correlation. A p-value of <0.05 is considered statistically significant correlation of the variables analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Bugude Shiva Shankar, MDS, Principal Investigator — College of Applied Health Sciences - Al Rass
Locations (1):
- Dr Bugude Shiva Shankar, Ar Rass, Al Qassim, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
The Research data will be available to the Principal Investigator. On requirement the data will be shared to whomsoever after consultation with the concerned higher authorities in the College of Applied Health sciences in Ar rass. The descriptive & analytical data will be used for scientific publication.